CLINICAL TRIAL: NCT03518151
Title: Women's Responses to Adjusted Product Placement and Its Effects on Diet - 1 (WRAPPED1)
Acronym: WRAPPED1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23361
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Diet Modification
Keywords: public health; dietary inequalities; environment design

STUDY DESIGN:
Intervention Model Description: WRAPPED1 is a natural experiment with a prospective matched controlled cluster design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention includes 3 components: i) creation of a new fresh fruit and vegetable section at store entrance; ii) placing frozen fruit and vegetables in the first aisle and iii) removal of all cakes, confectionary and sugar sweetened beverages from checkouts (replaced with non-food items, fruit and bottled water).
  Interventions: Other: Product placement intervention
- Control (Sham Comparator): The control condition is provision of a limited range of fresh fruit and vegetables, all placed at the back of the store, frozen vegetables in a middle aisle and confectionery sold at checkouts.
  Interventions: Other: Sham comparator

INTERVENTIONS:
Other: Product placement intervention — The intervention includes 3 components: i) creation of a new fresh fruit and vegetable section and island in the first aisle; ii) placing frozen fruit and vegetables in the first aisle and iii) removal of all cakes, confectionary and sugar sweetened beverages from checkouts (replaced with non-food items, fruit and bottled water).
  Arms: Intervention
Other: Sham comparator — The control condition is provision of a limited range of fresh fruit and vegetables, all placed at the back of the store, frozen vegetables in a middle aisle and confectionery sold at checkouts.
  Arms: Control

SUMMARY:
This research project aims to help address a gap in understanding about the micro-environmental determinants of diet by exploring whether improving the placement of fresh and frozen fruit and vegetables and removing temptations of confectionary at checkouts in discount supermarkets influences the dietary behaviours of women aged 18-45 years and whether it is cost effective.

DETAILED DESCRIPTION:
This study is a natural experiment with a prospective cluster controlled design. The intervention includes creating a new fresh fruit and vegetable section at the store entrance, placing frozen fruit and vegetable in the first aisle and removing confectionery from checkouts; it will be implemented continuously for 6 months in discount supermarkets.

The control condition is provision of a limited range of fresh fruit and vegetables, all placed at the back of the store, frozen vegetables in a middle aisle and confectionery sold at checkouts. Control and intervention stores will be located across England to improve generalizability of the sample. Each control store will be matched to an intervention store on i) sales profile, ii) customer profile and iii) neighbourhood deprivation (IMD deciles). Control stores will be located at least 50 miles from an intervention store to avoid contamination.

Women customers aged 18-45 years with a store loyalty card, who regularly shop at one of 3 intervention or 3 matched-control stores in England will be invited to participate. Women will be recruited via email, letter, SMS, shopping receipt note, Facebook advertisement, and in-store approach. Participants will contact the research team via text, email or Freephone and will be consented by phone after eligibility is assessed. Participants will be asked to complete four telephone surveys (baseline and 1, 3 and 6 months post intervention commencement) and will be offered 3x £10 Love2Shop vouchers that will be sent after completion of the baseline, 3 and 6 month surveys. A secure system to transfer store and participant loyalty card sales data has been established and confidentiality upheld through the use of study identification numbers.

Economic evaluation will be conducted from individual and retailer perspectives. Participant surveys will collect data about food expenditure, and travel costs to and from supermarkets that will be supplemented by loyalty card data. Refurbishment and ongoing costs, plus impact on sales will be estimated.

A process evaluation will be conducted to monitor intervention implementation (in-store surveys), mechanisms of impact (interviews with a sub-sample of supermarket staff and participants) and context (analysis of grocery shopping habits - location and frequency of different stores).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years
* Hold an store loyalty card
* Shop regularly in the 12-weeks before recruitment according to loyalty card data
* Shoppers who choose items in-store but opt for home delivery will be eligible

Exclusion Criteria:

* Women under the age of 18 or over 45 years
* Shopped less than once in 12-weeks prior to recruitment
* Online-only shopper
* No store loyalty card

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Dietary quality score | 3 month follow-up post intervention commencement
  The primary outcome is women's dietary quality measured using a 20-item food frequency questionnaire (FFQ) to create a standardised dietary quality score (validated against 100-item FFQ and red cell folate).

SECONDARY OUTCOMES:
Child's dietary quality score | 3 month follow-up post intervention commencement
  Child's dietary quality will be collected using a validated FFQ for use with parents of children aged 2-6 years.
Women's daily fruit and vegetable portions | 3 month follow-up post intervention commencement
  Women's daily fruit and vegetable portions will be collected using a 2-item tool that has been validated against urinary potassium and plasma ascorbic acid to describe high (≥5 portions/day) and low (≤2.5 portions/day) intake.
Women's weekly confectionery intake | 3 month follow-up post intervention commencement
  Frequency per week that women consume sweets and chocolates
Weekly sales of fresh fruit and vegetables | 12 week period following intervention commencement
  Total weekly sales of fresh fruit and vegetables collected via electronic sales data
Weekly sales of confectionery | 12 week period following intervention commencement
  Total weekly sales of confectionery collected via electronic sales data

REFERENCES:
- [Derived] Stuber JM, Beulens JW, Ayala GX, Crozier SR, Dijkstra SC, Lin SF, Vogel C, Mackenbach JD. Can nudge interventions targeting healthy food purchases in real-world grocery stores reduce diet-related health disparities? A pooled analysis of four controlled trials. Int J Behav Nutr Phys Act. 2024 Dec 3;21(1):137. doi: 10.1186/s12966-024-01687-3. PMID 39627771
- [Derived] Vogel C, Crozier S, Penn-Newman D, Ball K, Moon G, Lord J, Cooper C, Baird J. Altering product placement to create a healthier layout in supermarkets: Outcomes on store sales, customer purchasing, and diet in a prospective matched controlled cluster study. PLoS Med. 2021 Sep 7;18(9):e1003729. doi: 10.1371/journal.pmed.1003729. eCollection 2021 Sep. PMID 34491999